CLINICAL TRIAL: NCT00552591
Title: Family Heart Health Program: Randomized, Controlled Trial
Acronym: FHHP-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NA 6142
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Coronary Heart Disease
Keywords: family risk; behavior modification; lifestyle change; prevention of CHD; health care costs
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Family Heart Health Program
  Interventions: Behavioral: 12-week risk reduction program, managed by a Heart Health Educator
- 2 (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: 12-week risk reduction program, managed by a Heart Health Educator — The educator and participant will negotiate a personal plan for achieving the goals through lifestyle change (i.e. smoking cessation, increased exercise, improved nutrition) and, if necessary, pharmacotherapy coordinated by the participant's personal physician. Educational modules have been developed to address specific lifestyle issues including smoking cessation, healthy eating, exercise, and weight management, and will be provided to participants as required. A summary of the risk factor profile and personal plan will be incorporated into a report for the participant's personal physician as well. Participants will also receive telephone-based motivational counseling sessions for 12 weeks to address specific lifestyle issues.
  Arms: 1

SUMMARY:
Background: Family members (spouses, siblings, offspring) of patients with coronary heart disease (CHD) may themselves be at increased risk for developing CHD for genetic, biochemical and/or behavioural reasons. Targeted approaches aimed at family members of those with established CHD may be a cost-effective way to identify high-risk persons and link them to effective risk factor modification. During pilot testing we found 29% of family members of patients recently hospitalized at our institution had ≥ 3 CHD risk factors. Encouragingly, they indicated high levels of "readiness" to change underlying risk behaviours such as cigarette smoking and physical inactivity. We have developed a 12-week family heart health program featuring a personal plan for achieving risk factor goals and weekly contact with a heart health educator. This intervention needs to be fully tested.

Research Aims:

In this study, we will:

1. Compare the effects of a targeted family heart health (FHH) screening, counselling and follow-up program versus usual care (UC) for reducing participants total cholesterol/high density lipoprotein (TC/HDL) ratio 52 weeks after program entry, in family members of patients recently hospitalized with CHD;
2. Compare the effects of the FHH program versus UC on modifiable components comprising the Framingham score, including: smoking status; systolic blood pressure; total cholesterol; and high density lipoprotein cholesterol;
3. Compare the effects of the FHH program versus UC on: lifestyle-related factors (dietary patterns, leisure time exercise, body composition); medication use (anti-lipemic medications, anti-hypertensive medications, pharmacotherapies for smoking cessation); and use of healthcare resources (physician visits, hospitalization days, number of laboratory and diagnostic tests and procedures).

ELIGIBILITY:
Inclusion Criteria:

* Spouse, offspring or sibling of patient hospitalized at UOHI within the past 5 years for:

  1. Acute coronary syndrome (ACS);
  2. Elective percutaneous coronary intervention (PCI); or
  3. Bypass surgery (CABG);
* Willing to provide informed consent;
* At least one of the following modifiable risk factors:

  1. Current smoker;
  2. Systolic blood pressure ≥ 140 and or Diastolic BP ≥ 90 and/or currently on medication to treat high blood pressure;
  3. Total cholesterol/HDL-cholesterol ratio ≥ 5.0 and/or on antilipemic medication;
  4. Abdominal obesity (for men, waist circumference > 102 cm; for women, waist circumference > 88cm);
  5. Physical Inactivity [<150 min mod, 5-7 d/week or <100 min vig, 4-7 d/week]
* Geographically available for assessment, intervention and follow-up.

Exclusion Criteria:

1. Unable to understand English or French;
2. History of diabetes mellitus or any atherosclerotic disease;
3. Fasting glucose ≥ 7.0 mmol/L at screening;
4. Presence of life threatening illness (e.g., known or suspected cancer or other disease with a life expectancy of less than five years);
5. Chronic kidney disease and/or undergoing dialysis;
6. Active liver disease;
7. Pregnant or planning to become pregnant within the next year;
8. Cognitive impairment;
9. Other family member already participating in study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
TC/HDL ratio | one year

SECONDARY OUTCOMES:
Secondary outcomes of interest will include the modifiable components comprising the Framingham score (smoking status, systolic BP, total cholesterol, HDL- and LDL-cholesterol) | 12 weeks and one year
Use of risk reducing medications, use of health care resources, smoking status, leisure time exercise, dietary patterns, and body composition | 12 weeks and one year

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Reid, MBA, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation; Andrew L Pipe, MD, Study Chair — Ottawa Heart Institute Research Corporation; Lori J Mosca, MD, PhD, Study Chair — New York Presbyterian Hospital; Heidi Mochari, MPH, RD, Study Chair — New York Presbyterian Hospital; George Wells, PhD, Study Chair — Ottawa Heart Institute Research Corporation; Louise J Beaton, MSc, Study Chair — Ottawa Heart Institute Research Corporation; Pat O'Farrell, RN, Study Chair — Ottawa Heart Institute Research Corporation; Chris M Blanchard, PhD, Study Chair — Dalhousie University; Sophia Papadakis, MHA, Study Chair — Ottawa Heart Institute Research Corporation; Monika Slovinec D'Angelo, PhD, Study Chair — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Reid RD, McDonnell LA, Riley DL, Mark AE, Mosca L, Beaton L, Papadakis S, Blanchard CM, Mochari-Greenberger H, O'Farrell P, Wells GA, Slovinec D'Angelo ME, Pipe AL. Effect of an intervention to improve the cardiovascular health of family members of patients with coronary artery disease: a randomized trial. CMAJ. 2014 Jan 7;186(1):23-30. doi: 10.1503/cmaj.130550. Epub 2013 Nov 18. PMID 24246588